CLINICAL TRIAL: NCT07262775
Title: Radicle Relief RAL™: A Randomized, Double-Blind, Placebo-Controlled Study Assessing the Impact of Health and Wellness Products on Pain Relief and Related Health Outcomes
Brief Title: Radicle Relief RAL™: A Study Assessing the Impact of Health and Wellness Products on Pain Relief and Related Health Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX_P_2503_RAL
Record Dates: First submitted 2025-11-18; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Pain Interference

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on their assigned sex at birth and health outcome score during enrollment, then randomized to one of the study arms. Each participant will have an equal chance of being assigned to any study arm.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Control (Placebo Comparator): Pain Relief Supplement Product Placebo Control
  Interventions: Dietary Supplement: Pain Relief Supplement Product Placebo Control
- Active Relief Product 1 (Experimental): Pain Relief Supplement Active Product 1
  Interventions: Dietary Supplement: Pain Relief Supplement Active Product 1

INTERVENTIONS:
Dietary Supplement: Pain Relief Supplement Product Placebo Control — Participants will use their Pain Relief Supplement Product Placebo Control as directed for a period of 8 weeks
  Arms: Placebo Control
Dietary Supplement: Pain Relief Supplement Active Product 1 — Participants will use their Pain Relief Supplement Active Product 1 as directed for a period of 8 weeks
  Arms: Active Relief Product 1

SUMMARY:
Radicle Relief RAL: A randomized, double-blind, placebo-controlled study assessing the impact of health and wellness products on pain relief and related health outcomes.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants will (1) have the opportunity for meaningful improvement (at least 30%) in their primary health outcome, and (2) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 8 weeks. Participant reports of health indicators will be collected at enrollment and throughout the active period of study product usage. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
3.1 Inclusion

Participants must meet all the following criteria:

* Adults, at least 21 years of age at the time of electronic consent, inclusive of all ethnicities, races, and gender identities

  * Assigned sex at birth will determine sex-specific recruitment and surveys (male vs female) employed, when needed
* Resides in the United States
* Has the opportunity for at least 30% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

3.2 Exclusion

Individuals who report any of the following during screening may be excluded from participation:

* Report being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English at a 7th grade level
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients.

  * NYHA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients.

  * Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOIs, or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study products and/or pose a safety risk
* Lack of reliable daily access to the internet

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 715 (Estimated)
Dates: Start 2026-01-04 (Estimated); Primary Completion 2027-01-04 (Estimated); Study Completion 2027-01-04 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Interference | 9 weeks
  Change in Pain Interference: Difference in rates of change over time in pain interference score as assessed by PROMIS Pain Interference 6A (scale 6-30; with higher scores corresponding to more severe pain interference)

SECONDARY OUTCOMES:
Change in Pain Intensity | 9 weeks
  Change in Pain Intensity: Difference in rates of change over time in pain intensity score as assessed by PROMIS Pain Intensity 3A (scale 3-15; with higher scores corresponding to more severe pain intensity)
Change in sleep | 9 weeks
  Change in sleep: Difference in rates of change over time in sleep score as assessed by PROMIS Sleep Disturbance 8A (scale 8-40; where higher scores correspond to higher levels of sleep disturbance)
Change in Physical Function | 9 weeks
  Change in physical function: Difference in rates of change over time in physical function score as assessed by Patient Reported Outcome Measurement System (PROMIS) Physical Function 8C (scale 8-40; where higher scores correspond to better physical function)

OTHER OUTCOMES:
Minimal clinically important difference (MCID) in pain interference | 9 weeks
  Minimal clinically important difference (MCID) in pain interference: Likelihood of experiencing minimal clinically important difference in pain interference, as measured by PROMIS Pain interference (6-30; where lower scores indicate less pain interference).
Minimal clinically important difference (MCID) in pain intensity | 9 weeks
  Minimal clinically important difference (MCID) in pain intensity: Likelihood of experiencing minimal clinically important difference in pain intensity, as assessed by PROMIS Pain Intensity 3A (scale 3-15; with higher scores corresponding to more severe pain intensity)
Minimal clinically important difference (MCID) in sleep | 9 weeks
  Minimal clinically important difference (MCID) in sleep: Likelihood of experiencing minimal clinically important difference in sleep score as assessed by PROMIS Sleep Disturbance 8A (scale 8-40; where higher scores correspond to higher levels of sleep disturbance)
Minimal clinically important difference (MCID) in Physical Function | 9 weeks
  Minimal clinically important difference (MCID) in physical function: Likelihood of experiencing minimal clinically important difference in physical function score as assessed by PROMIS Physical Function 8C (scale 8-40; where higher scores correspond to better physical function)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hewlings, Principal Investigator — Radicle Science
Locations (1):
- Radicle Science Inc., Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Related Info — https://www.radiclescience.com